CLINICAL TRIAL: NCT05171933
Title: Educational Status, Stress Factors and Vaccine Attitudes Among Dental Students During COVID-19 Pandemic in Turkey
Brief Title: Stress Factors and Vaccine Attitudes Among Dental Students During COVID-19
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Dilber Bilgili Can, Assistant Professor, Yuzuncu Yil University
Other Study IDs: 2021/04-13
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Surveys and Questionnaires
Keywords: COVID-19; vaccine; anxiety; concern; dental students
MeSH Terms: conditions — COVID-19; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — This study is based on a survey made on COVID-19

SUMMARY:
Background: The aim of this study is to investigate the impact of the COVID-19 pandemic on the education of dental students in Turkey, the reasons that affect the psychological attitudes of students towards this disease, stress factors and the effect of these factors on vaccine acceptance.

Methods: The survey was applied online and consisted of questions aimed to find out the demographic characteristics, educational status, anxiety-stress factors, and reasons for students' decision behind COVID-19 vaccine administration. The psychological impact of COVID-19 was assessed by means of the Generalised Anxiety Disorder-7 scale (GAD-7). Standard descriptive statistics, the chi-square test and independent samples t test were used for statistical analysis.

DETAILED DESCRIPTION:
An online survey was conducted among dentistry students in Turkey between April-May 2021. Participants were included in the survey on the condition that they were enrolled in a dental school in Turkey at the time.

Participation in the survey was completely voluntary. Participants got the link to the survey online and accessed it directly by clicking the link. At the beginning of the survey, participants were informed that their participation was voluntary, their answers were anonymous, and they could leave at any time. They were then explicitly asked if they wanted to participate in the research study before starting the survey. The survey was created using the free-to-access Google Forms app and took approximately 15 minutes to complete.

Survey consisted of questions about the effects of COVID-19 epidemic on the education of dental students in Turkey, stress factors, the reasons and factors affecting their psychological attitudes towards this disease. There were also questions about the effects of these reasons/factors on attitudes and behaviors related to vaccination.

ELIGIBILITY:
Inclusion Criteria: To be a dental student in Turkey -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dental studentS in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Educational Status, Stress Factors and Vaccine Attitudes among Dental Students during COVID-19 Pandemic in Turkey | April-May 2021
  The aim of this study is to investigate the impact of the COVID-19 pandemic on the education of dental students in Turkey, the reasons that affect the psychological attitudes of students towards this disease, stress factors and the effect of these factors on vaccine acceptance.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No